CLINICAL TRIAL: NCT01548950
Title: Combined Clinical and Surgical Approaches to Congenital Heart Disease Associated With Pulmonary Arterial Hypertension (PAH-CHD)
Brief Title: Drug Therapy and Surgery in Congenital Heart Disease With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto do Coracao (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPPesq 0502/11
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2015-06

CONDITIONS: Congenital Heart Disease; Pulmonary Arterial Hypertension
Keywords: Congenital heart disease; Pulmonary arterial hypertension; Sildenafil; Bosentan; Pediatric cardiac surgery
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm study (Other): Preoperatively, sildenafil until development of pulmonary congestion (1-4 weeks). On treatment pulmonary congestion (dyspnea and need for increasing diuretics) occurs when there is a substantial decrease in pulmonary vascular resistance, which may be confirmed noninvasively by Doppler-echocardiography. At that moment, patient will be assigned to surgery. If pulmonary congestion is not observed, bosentan will be added on top of sildenafil, and the patient will be kept on treatment for 10-12 months. In this case, a new cardiac catheterization will be performed before surgery. In both cases (short-term and medium-term treatment) patients will be kept on treatment for six months following surgery, and then re-catheterized.
  Interventions: Drug: Sildenafil singly or in association with Bosentan

INTERVENTIONS:
Drug: Sildenafil singly or in association with Bosentan — Sildenafil, 1-4 mg/Kg/day (6-hour intervals) preoperatively, until development of pulmonary congestion (generally 1-4 weeks) or preoperatively, for 10-12 months, in association with bosentan (15.6-62.5 mg b.i.d.) if pulmonary congestion does not develop. Surgery will be performed at 1-4 weeks (short-term treatment) or at 10-12 months (medium-term treatment) if operability criteria are met (catheterization). In both cases (short and medium-term treatments), the drug or drugs will be kept for 6 months postoperatively, when final catheterization will be performed for efficacy testing.

SUMMARY:
The purpose of this study is to test the hypothesis that treating PAH-CHD patients preoperatively with PAH drugs and keeping them on treatment for six months after surgery reduces the risk of immediate postoperative death and the risk of residual PAH at six months following operation to <10%.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a complicating factor in the management of congenital heart disease (CHD) with intracardiac or extracardiac communications. In children with moderate to severe PAH, the risk of serious complications following the surgical repair of shunts (including right cardiac failure and death) is 15-20% or even higher, and the risk of late, postoperative residual PAH is ~25%. We therefore intend to conduct a study aimed at reducing the risk of severe immediate postoperative complications and the risk of residual PAH at six months following surgery to less than 10% in children with moderate PAH (primary objective). The study is also aimed at promoting a statistically significant reduction in pulmonary artery pressure and pulmonary vascular resistance at six month after surgery, compared with baseline in children with moderate or severe PAH (secondary objective). We hypothesized that these goals could be achieved by treating patients preoperatively and for six months postoperatively with sildenafil, either singly or combined with bosentan. Both drugs have been approved for treatment of PAH on the basis of randomized clinical trials. Preoperative and postoperative (on treatment) hemodynamic evaluation will be based on noninvasive and invasive diagnostic procedures. As an additional objective, we intend to analyze possible abnormalities in genes that have been shown to be associated with PAH-CHD, and inflammatory mediators as well. The idea is to investigate whether changes in these markers correlate with the clinical profile and response to treatments.

ELIGIBILITY:
Inclusion Criteria:

* Potentially operable patients with congenital cardiac septal defects (bi-ventricular physiology) and PAH, must have at least three of the following severity criteria: age > 18 months; absence of congestive heart failure (pulmonary congestion); Down syndrome; bidirectional shunting across the septal defect; periods of systemic (peripheral) oxygen saturation < 90%.

Exclusion Criteria:

* Patients with complex cardiac anomalies for whom there are no possibilities of complete repair. Patients with uni-ventricular physiology.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Immediate postoperative right cardiac failure and mortality, and prevalence of residual PAH six months after surgery. | Six months following surgery
  Drug treatment must reduce the prevalence of immediate postoperative right cardiac failure / death to <10%, and the prevalence of residual PAH six months after cardiac surgery to <10%. Residual PAH is defined as an elevation of mean pulmonary artery pressure above 25 mmHg, and elevation of pulmonary vascular resistance above 3.0 Wood units x squared meters (body surface area).

SECONDARY OUTCOMES:
Pulmonary vascular resistance six months after surgical repair of congenital cardiac shunts with PAH | Six months following surgery
  Drug treatment before surgery and maintained for six months following repair of congenital cardiac shunts must promote a statistically significant reduction in pulmonary vascular resistance (at six months) compared with baseline (preoperative) level.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Augusto Lopes, M.D., Principal Investigator — Instituto do Coração (InCor) - HCFMUSP - São Paulo - Brazil
Locations (1):
- Instituto do Coração (InCor) HCFMUSP, São Paulo, Brazil